CLINICAL TRIAL: NCT02108210
Title: Cytokine Inhibition in Chronic Fatigue Syndrome Patients
Acronym: CiCFS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R0002198; 2013-005466-19 (EudraCT Number); NL47571.091.14 (Other: Toetsingonline)
Record Dates: First submitted 2014-03-21; First posted 2014-04-09 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic fatigue syndrome; Cytokines; Interleukin-1; Fatigue; Anakinra
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anakinra (Experimental): This therapy will consist of once daily subcutaneous injections (100mg/day) during a period of 4 weeks. Patients will be monitored at week 1 and week 4 after starting medication for development of side effects. Therapy will be stopped in case of severe side effects, interfering disease or pregnancy. During the intervention period, use of co-medication is only allowed when used for ≤14 consecutive days, on the condition that there are no known interactions with anakinra. Oral contraceptives and/or paracetamol can be used without a limitation. During the follow-up period, there are no limitations regarding the use of medication. All co-medication will be registered precisely and reported afterwards.
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Patients in the placebo group will also receive once daily subcutaneous injection during a period of 4 weeks. Placebo injections will be identically in appearance compared to the Anakinra injections. Patients in the placebo group will have the same visits and monitoring for side effects as the patients randomized to the other treatment arm.
  During the intervention period, use of co-medication is only allowed when used for ≤14 consecutive days, on the condition that there are no known interactions with anakinra. Oral contraceptives and/or paracetamol can be used without a limitation. During the follow-up period, there are no limitations regarding the use of medication. All co-medication will be registered precisely and reported afterwards.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo
  Arms: Placebo

SUMMARY:
Rationale: Chronic fatigue syndrome (CFS) is a medically unexplained syndrome for which no somatic or pharmacological treatment has been proven effective. Dysfunction of the cytokine network has been suspected to play a role in the pathophysiology of CFS. Although derangements of the cytokine network in CFS are controversial, a major problem is that many studies did not use adequate controls. In addition, all studies have been performed on peripheral venous blood of the patients. As cytokines mainly act in the tissues, e.g., the brain, the information that can be derived from peripheral blood cells is limited. The only information regarding the possible role of cytokines in the pathophysiology of CFS could come from intervention studies in which pathogenetically important cytokines are inhibited. A potentially relevant cytokine which can be blocked in humans without severe side effects is IL-1. Although it is plausible that these cytokines play a role in CFS, there is limited evidence for this.

Objective: To investigate the effect on symptomatology of interference with IL-1 in CFS patients.

Study design: A randomized placebo controlled study will be performed to determine whether interference with IL-1 is able to reduce fatigue and disabilities in CFS patients.

Study population: Female CFS patients without psychiatric co-morbidity will be included in this study. Patients of the outpatient clinic of the Department of General internal medicine and the Expert Centre for Chronic Fatigue (ECCF) will be asked to participate in the study. Patients will be asked to bring a healthy neighbourhood control to their first study visit.

Intervention: After inclusion patients will be randomized to receive one of the following treatments:

* interleukin-1 inhibitor Anakinra (IL-1Ra) for 4 weeks (N=25);
* placebo for 4 weeks (N=25).

Main study parameters/endpoints: The primary outcome measure will be fatigue severity measured with the Checklist Individual Strength (CIS) at 4 weeks, measurement will be repeated up to 26 weeks.

Secondary outcome measures will be:

* level of functional impairment measured with the Sickness Impact Profile (SIP8) total score;
* physical and social functioning assessed with the subscale physical functioning and social functioning of the SF-36;
* level of psychological distress assessed with the total score on the Symptom Checklist-90 (SCL-90);
* pain severity assessed with a Visual Analog Scale (VAS);
* cytokine measurement in blood (plasma and blood in Pax-gene tubes) and saliva (at protein and mRNA level);
* cortisol measurement in saliva and hair;
* microbiome determination in faeces;
* body temperature and pulse rate.

ELIGIBILITY:
Inclusion Criteria:

* CDC-diagnosed CFS-patients;
* female, between 18 and 59 years old;
* fatigue duration ≤10 years, or significant increase of complaints during the last 10 years
* score of ≥40 on the subscale fatigue severity of the CIS (Checklist Individual Strength);
* marked functional impairment assessed with the Sickness Impact Profile (SIP-8) and operationalised as a total score of ≥700.

Exclusion Criteria:

* pregnant or nursing women;
* women who intend to get pregnant during the study;
* fatigue duration >10 years;
* patients who use or have used psychotropic medication in the past month;
* substance abuse in the past 3 months;
* patients taking any medication except oral contraceptives and/or paracetamol;
* patients with evident somatic co-morbidity;
* previous or current engagement in CFS research;
* inability to understand the nature and the extent of the trial and the procedure required;
* psychiatric co-morbidity (major depression, psychosis, eating disorders, anxiety disorders, bipolar disease and post traumatic stress disorder) assessed with the MINI;
* live vaccination during the past four weeks;
* current engagement in a legal procedure with respect to disability claims.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
CIS (checklist individual strength, compared to baseline) | 4 weeks, measurement will be repeated up to 26 weeks
  To investigate the role of the cytokine IL-1 in the pathogenesis of CFS and to find leads for future treatment of CFS, a disorder for which there is no proven effective drug treatment. The primary outcome measure will be fatigue severity at 4 weeks measured with the Checklist Individual Strength (CIS).

SECONDARY OUTCOMES:
SIP8 (sickness impact profile, change from baseline) | 4 weeks, measurement will be repeated up to 26 weeks
  level of functional impairment
SF-36 (subscale physical functioning and social functioning, compared to baseline) | 4 weeks, measurement will be repeated up to 26 weeks
  physical and social functioning assessed with the subscale physical functioning and social functioning of the SF-36
SCL-90 (symptom checklist-90, compared to baseline) | 4 weeks, measurement will be repeated up to 26 weeks
  level of psychological distress assessed with the total score on the Symptom Checklist-90
VAS pain (visual analog scale, compared to baseline) | 4 weeks, measurement will be repeated up to 26 weeks
  pain severity assessed with a Visual Analog Scale
Cortisol in saliva and hair (concentration compared to baseline) | 4 weeks
  Because of the possible role of the hypothalamus-pituitary-adrenal axis we will also measure the cortisol concentration in saliva and hair. For the baseline assessment, comparison will be made with matched neighbourhood controls.
microbiome determination faeces | at baseline
  A new field of great interest in pathophysiology is the role of the microbial flora of the host (microbiome). The availability of well defined patients with CFS and matched controls is a great opportunity in an unexplored area of CFS research, to assess whether the microbiome of CFS patients is peculiar.
cytokine concentrations in blood and saliva (compared to baseline) | 4 weeks
  In addition to the cytokine intervention, we will assess cytokines (at the transcriptional level and as proteins) in serum and saliva at baseline and after 4 weeks of intervention. For the baseline assessment, comparison will be made with matched neighbourhood controls.

OTHER OUTCOMES:
Body temperature | 4 weeks, measurement will be repeated up to 26 weeks
pulse rate | 4 weeks, measurement will be repeated up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jos van der Meer, Prof, PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Roerink ME, Knoop H, Bronkhorst EM, Mouthaan HA, Hawinkels LJAC, Joosten LAB, van der Meer JWM. Cytokine signatures in chronic fatigue syndrome patients: a Case Control Study and the effect of anakinra treatment. J Transl Med. 2017 Dec 29;15(1):267. doi: 10.1186/s12967-017-1371-9. PMID 29284500
- [Derived] Roerink ME, Bredie SJH, Heijnen M, Dinarello CA, Knoop H, Van der Meer JWM. Cytokine Inhibition in Patients With Chronic Fatigue Syndrome: A Randomized Trial. Ann Intern Med. 2017 Apr 18;166(8):557-564. doi: 10.7326/M16-2391. Epub 2017 Mar 7. PMID 28265678
- [Derived] Roerink ME, Knoop H, Bredie SJ, Heijnen M, Joosten LA, Netea MG, Dinarello CA, van der Meer JW. Cytokine inhibition in chronic fatigue syndrome patients: study protocol for a randomized controlled trial. Trials. 2015 Oct 5;16:439. doi: 10.1186/s13063-015-0971-z. PMID 26438161